CLINICAL TRIAL: NCT02295384
Title: Use of Concomitant Medications in HIV-1 Infected Patients in a Large Community Practice in Sydney, Australia
Status: Completed | Type: Observational
Sponsor: Holdsworth House Medical Practice (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Principal Investigator, Dr. Mark Bloch, Principle Investigator, Holdsworth House Medical Practice
Other Study IDs: Polypharmacy Audit
Record Dates: First submitted 2014-11-17; First posted 2014-11-20 (Estimated); Last update posted 2016-09-12 (Estimated); Status verified 2016-09

CONDITIONS: HIV
Keywords: Polypharmacy; Medication Therapy Management

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Audit Group: Patients attending HHMP in Darlinghurst, Sydney, New South Wales with documented HIV-1 infection from 1st January 2005 to 31st July 2014, who were considered "linked to care" (Attendance during the study period for at least 2 visits >3 months and <12 months apart with measured laboratory virological or immunological markers (either on-site or at a co-management site)).
  Interventions: Other: Retrospective Audit

INTERVENTIONS:
Other: Retrospective Audit — Retrospective Audit

SUMMARY:
For the majority of patients, management of HIV-1 infection involves effective and well tolerated antiretroviral therapy with simplified pill load and dosing, exemplified by the availability of single tablet regimens (STRs) with single tablet once daily dosing. STR therapy has been shown to improve adherence and reduce hospitalisations (Cohen et al., 2013; Sax et al., 2012).

However, the aging of the HIV cohort in Australia and globally has raised issues of increasing co-morbidities and consequent polypharmacy to manage these (Jansson & Wilson, 2012; Edelman et al., 2013).

Polypharmacy may not only impact on adherence, but also increases the potential for drug-drug interactions (Holtzman et al., 2013).

Stribild, a highly effective STR, contains cobicistat to boost the levels of the component integrase inhibitor, elvitegravir. Cobicistat does not have antiretroviral activity, but acts by inhibiting Cyp3A4 of the cytochrome p450 metabolic pathway. Other drugs metabolized via this pathway may be affected by this drug-drug interaction (Rogatto et al., 2014). Additionally there is evidence of increased risk of nephrotoxicity with co-administration of tenofovir and non-steroidal anti-inflammatory medication (NSAIDS) (Marcotte et al., 2008).

Data on use of concomitant medications in Australian patients with HIV is sparse. This study aims to determine, in a large caseload community HIV practice, the use of concomitant medications in HIV, patient pill load and dosing frequency, and potential drug-drug interactions with stribild.

ELIGIBILITY:
Inclusion Criteria:

* Documented HIV-1 infection
* Attendance during the study period for at least 2 visits >3 months and <12 months apart with measured laboratory virological or immunological markers (either on-site or at a co-management site).

Exclusion Criteria:

* Attendance by patient with HIV infection who does not have laboratory markers of HIV viral load or CD4 count
* Incomplete/inaccessible patient records

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV-infected patients attending HHMP from 1st January 2005 to 31st July 2014 inclusive, who had at least 2 practice visits separated by ≥90 days in a year involving HIV laboratory monitoring whilst attending HHMP (either on-site or at a co-management site).
Sampling Method: Non-Probability Sample
Enrollment: 1104 (Actual)
Dates: Start 2014-11; Primary Completion 2015-12 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Quantity of concomitant medications used in patients with HIV-1 infection | 9.5 years
  The pill burden of concomitant medications for patients with HIV-1 infection
Types of concomitant medications used in patients with HIV-1 infection | 9.5 years

SECONDARY OUTCOMES:
Total pill load in patients with HIV | 9.5 years
Frequency of drug dosing | 9.5 years
Use of concomitant medications that could have potential drug-drug interaction with stribild (co-formulated elvitegravir/cobicistat/tenofovir/emtricitabine) | 9.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Mark Bloch, MBBS, M Med, Principal Investigator — Holdsworth House Medical Practice
Locations (1):
- Holdsworth House Medical Practice, Darlinghurst, New South Wales, Australia

REFERENCES:
- [Background] Jansson J, Wilson DP. Projected demographic profile of people living with HIV in Australia: planning for an older generation. PLoS One. 2012;7(8):e38334. doi: 10.1371/journal.pone.0038334. Epub 2012 Aug 9. PMID 22912660
- [Background] Edelman EJ, Gordon KS, Glover J, McNicholl IR, Fiellin DA, Justice AC. The next therapeutic challenge in HIV: polypharmacy. Drugs Aging. 2013 Aug;30(8):613-28. doi: 10.1007/s40266-013-0093-9. PMID 23740523
- [Background] Holtzman C, Armon C, Tedaldi E, Chmiel JS, Buchacz K, Wood K, Brooks JT; , and the HOPS Investigators. Polypharmacy and risk of antiretroviral drug interactions among the aging HIV-infected population. J Gen Intern Med. 2013 Oct;28(10):1302-10. doi: 10.1007/s11606-013-2449-6. Epub 2013 Apr 20. PMID 23605401
- [Result] Cohen CJ, Meyers JL, Davis KL. Association between daily antiretroviral pill burden and treatment adherence, hospitalisation risk, and other healthcare utilisation and costs in a US medicaid population with HIV. BMJ Open. 2013 Aug 1;3(8):e003028. doi: 10.1136/bmjopen-2013-003028. PMID 23906955
- [Result] Sax PE, Meyers JL, Mugavero M, Davis KL. Adherence to antiretroviral treatment and correlation with risk of hospitalization among commercially insured HIV patients in the United States. PLoS One. 2012;7(2):e31591. doi: 10.1371/journal.pone.0031591. Epub 2012 Feb 24. PMID 22384040
- [Result] Bpharm SM, Talbot A, Trottier B. Acute renal failure in four HIV-infected patients: Potential association with tenofovir and nonsteroidal anti-inflammatory drugs. Can J Infect Dis Med Microbiol. 2008 Jan;19(1):75-6. doi: 10.1155/2008/370535. No abstract available. PMID 19145267
- See also: Co-prescription of Non-HIV Medications in HIV-Infected Individuals in 5 European Countries and the Possible Impact of Interactions With Elvitegravir/Cobicistat/Emtricitabine/Tenofovir (E/C/F/TDF) — http://www.hiv-druginteractions.org/data/NewsItem/115_15_PKW_HIV.pdf